CLINICAL TRIAL: NCT01350713
Title: Testing the Counter-irritating Efficacy of Topical Povidone-iodine in Thermal Burns; Comparison to Conventional Treatments
Brief Title: The Counter-irritating Efficacy of Topical Povidone-iodine in Thermal Burns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Arie Bahir, Sherute Briut Clalit ( HMO)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 060/2011K
Record Dates: First submitted 2011-05-08; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2011-05

CONDITIONS: Skin Burns
Keywords: skin; burn; povidone iodine; cold water
MeSH Terms: conditions — Paresthesia; Burns | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- povidone iodine (Experimental)
  Interventions: Drug: povidone iodine
- cold water (Active Comparator): treatment by cold water after burn
  Interventions: Drug: povidone iodine

INTERVENTIONS:
Drug: povidone iodine — one local application of 10% povidone iodine ointment
  Other Names: polydine ointment

SUMMARY:
Skin burns are one of the causes of disability, suffering and death in humans. Anecdotal, uncontrolled studies have shown the efficacy of povidone-iodine ointment in human skin burns, provided the preparation was applied shortly after the exposure to the heat source. The proposed study will conduct a controlled study in which the effect of povidone-iodine ointment will be tested in large group of patients and will be compared with standard cold water treatment.

DETAILED DESCRIPTION:
Skin burns are one of the causes of disability, suffering and death in humans. The current treatment includes application of cold water or other plant origin preparations. However non of these treatments was shown to be efficacious.

Animal studies have demonstrated the pronounced protective effect of povidone-iodine ointment against thermal burns. Moreover, anecdotal, uncontrolled studies in humans have shown the efficacy of povidone-iodine ointment in human skin burns, provided the preparation was applied shortly after the exposure to the heat source. The proposed study will conduct a controlled study in which the effect of povidone-iodine ointment will be tested in large group of patients and will be compared with standard cold water treatment.

ELIGIBILITY:
Inclusion Criteria:

* skin burns in children

Exclusion Criteria:

* allergy to iodine

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 280 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
prevention of skin lesions caused by exposure to heat source | 1 year
  Skin exposed to hot liquid or metal that topically treated with povidone-iodine will show no or slight irritation while individuals treated with the standard cold water will show strong skin irritation including erythema and blisters.

SECONDARY OUTCOMES:
scar prevention | 1 year
  povidine treated individuals no scar will develop. standard cold water treated patients may develop skin lesions(scars)

CONTACTS AND LOCATIONS:
Overall Officials: Arieh Bahir, MD, Principal Investigator — Sherute Briut Clalit
Locations (1):
- Sherute Briut Clalit, Tel Aviv Region, Gush Dan, Heifa, Beer Sheva, Israel